CLINICAL TRIAL: NCT07281534
Title: Analysing the Test-Retest Reliability of Cardiopulmonary Exercise Testing With Echocardiography
Brief Title: Test-Retest Reliability of Cardiopulmonary Exercise Testing With Echocardiography
Acronym: REPEATCPETecho
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Z-2024011
Record Dates: First submitted 2024-02-26; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Dyspnea; Cardiac
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Repeat CPET echo with a one-week interval
  Interventions: Diagnostic Test: CPETecho

INTERVENTIONS:
Diagnostic Test: CPETecho — repeat CPETecho with a one-week interval

SUMMARY:
CPETecho is progressively employed in diagnostic settings for pathophysiological detection, offering comprehensive assessment of both pulmonary and cardiac functions. This technique evolves from its invasive counterpart, where a diagnostic catheter is employed for hemodynamic monitoring, by substituting the invasive component with non-invasive echocardiography. Nevertheless, data on the test-retest reliability of CPETecho remain sparse, a factor critical in differentiating between measurement effects and actual therapeutic impacts.

ELIGIBILITY:
Inclusion Criteria:

* Capable of performing a maximal exercise test.
* Provide signed and dated informed consent.

Exclusion Criteria:

- Unstable symptoms, whereby therapy cannot be delayed for a week.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient (ICC) | Up to 2 weeks
  Analysing the Test-Retest Reliability of Cardiopulmonary Exercise Testing with Echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No